CLINICAL TRIAL: NCT02507999
Title: Goal-directed Therapy in Endovascular Coiling of Cerebral Aneurysm Patients - A Prospective, Blinded Randomized Controlled Trial
Brief Title: Goal-directed Therapy in Endovascular Coiling of Cerebral Aneurysm Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Jason Chui, Anesthetist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GDT
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal Directed Therapy - Flotrac Use Arm (Experimental): This arm will employ the use of the Flotrac device to monitor cardiac output, cardiac index, stroke volume, stroke volume variation, and blood pressure management.
  Interventions: Device: Flotrac
- Non-Goal Directed Therapy (No Intervention): In this arm, patients will have the Flotrac machine attached to their arterial catheter but the screen that displays the monitor readings will be covered and machine alarms will be turned off. The anesthesiologist will not be aware of the Flotrac monitor readings.

INTERVENTIONS:
Device: Flotrac — Flotrac guided intervention
  Arms: Goal Directed Therapy - Flotrac Use Arm

SUMMARY:
Goal directed therapy (GDT) is a technique, which employs a non-invasive cardiac output monitoring (NICOM) device to guide management of circulating blood volume and blood pressure during procedures. The purpose of this study is to determine whether the use of goal-directed therapy to optimize blood volume and cardiac output during the procedure can improve the outcome of patients undergoing endovascular treatment of a brain aneurysm.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) as a result of ruptured intracranial cerebral aneurysms is a life threatening condition; with an estimated incidence of 6-10 cases per 100,000 persons per year. Endovascular coil emobolization of the aneurysm is performed to isolate the aneurysm and reduce the risk of re-bleeding. Unfortunately, despite timely and successful intervention approximate 25% of post-coiling patients suffer immediate and/or long-term injury including death as a result of intracranial bleeding. This is mainly a consequence of subarachnoid hemorrhage-related complications , especially cerebral vasospasm. Angiographic vasospasm and symptomatic vasospasm occur in 30-70% and 20-30% of SAH patients respectively. Goal-directed therapy (GDT) provides a means to assess and manage circulating volume and cardiac output. In this study, the investigators would investigate the use of GDT during aneurysm coiling procedures can improve the clinical course of these patients.

This will be a blinded, randomized pilot study to compare clinical outcomes for endovascular coiling patients allocated to one of two treatments: GDT or non-GDT. Randomization consented patients will be randomized into GDT or non-GDT groups in 1:1 ratio. The attending anesthesiologists will not be blinded because of the nature of the intervention. However, surgeons, patients, outcomes assessors will be blinded as to the treatment intervention.

In all patients, an arterial catheter (routinely used in these patients) will be inserted and connected to the Flotrac (Edward Lifesciences). After transferring the patients into the angiogram suite, routine monitoring such as pulse oximetry, electrocardiography, non-invasive blood pressure monitoring, end-tidal CO2 and temperature probe will be attached to the patients. Anesthesia will be conducted in the standard fashion. Patients will be randomized into two groups in 1:1 ratio: GDT or non-GDT therapy.

* GDT group: the attending anesthesiologist will use the data obtained from the Flotrac to manage fluid and hemodynamics during the procedure following the prescribed treatment algorithm. The treatment interventions will start on induction of anesthesia and continue until the patients are extubated or transferred back to intensive care unit with mechanical ventilation.
* Non-GDT group: Flotrac will be connected but the machine values will be blinded to the anesthesiologist and interventionist. The screens of the Flotrac will be covered by opaque plastic bag and the alarms will be turned off. The attending anesthesiologist will make clinical decisions regarding the management of fluids and hemodynamics based on current individual routine practices.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age> 18 years of age) scheduled for aneurysm endovascular coiling procedures over the next 2 years.
* Grade I to IV SAH within 5 days of presentation will be included in the study.
* Only patients identified as appropriate by the neurosurgeon/neuro-radiologist will be recruited.

Exclusion Criteria:

- Patients with un-ruptured aneurysm(s)

* Patients with previous clipping or coiling procedure for the same aneurysm.
* Patients undergoing concomitant extracranial-intracranial bypass procedures or other non-neurosurgical procedures.
* Patients with giant aneurysm (size> 25mm)
* Pediatric patients (<18 years of age) or pregnant patients
* Unable to obtain informed consent from patients or substitute decision maker (SDM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Composite outcomes of cerebral vasospasm, stroke and death | 30 days
  To determine if the use of the Flotrac device during surgery is able to decrease the morbidity and mortality rates for 30 days following surgery

SECONDARY OUTCOMES:
Composite outcomes of all perioperative complications | 7 days, 30 days, 90 days
  To assess the rate of occurrence of neurological and cardiopulmonary complications that may arise up to 90 days following the participant's surgical procedure. This will be assessed at 7 days, 30 days, and 90 days from the point of study entry.
Neurological outcomes | 7 days, 30 days, 90 days
  Incidence of poor functional neurological outcomes at 7 days, 30 days and 90 days after the procedures.
Length of hospital stay | From study entry until hospital discharge, or up to 90 days of after the procedure
  Total length of stay in the neuro-critical care unit and in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MBChB, Principal Investigator — Assistant Professor, Western Unviersity
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No